CLINICAL TRIAL: NCT05601778
Title: Phase 2 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of HSK31858 in Participants with Non-cystic Fibrosis Bronchiectasis
Brief Title: A Study of HSK31858 in Participants with Non-Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK31858-201
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Non-cystic Fibrosis Bronchiectasis (NCFBE)
Keywords: HSK31858; NCFBE; phase II

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HSK31858 20mg (Experimental): multiple oral doses: 20mg/d for 24w
  Interventions: Drug: HSK31858
- HSK31858 40mg (Experimental): multiple oral doses: 20mg/d for 24w
  Interventions: Drug: HSK31858
- placebo (Placebo Comparator): multiple oral doses for 24w
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HSK31858 — HSK31858 is a novel inhibitor of DPP1 developed by Hisco Pharmaceutical and can reduce pulmonary exacerbations over a 24-week treatment period in patients with non-cystic fibrosis bronchiectasis
  Arms: HSK31858 20mg; HSK31858 40mg
Drug: placebo — the placebo comparator of study
  Arms: placebo

SUMMARY:
This is a phase II, randomised, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of HSK31858 in non-cystic fibrosis bronchiectasis (NCFBE) participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years and BMI≥18.0 kg/m^2 at the time of signing the ICF.

  2. Chest HRCT showed bronchiectasis affecting one or more lobes and was confirmed by a clinician as NCFBE(clinically characterized by chronic cough, expectoration and/or intermittent hemoptysis, with or without shortness of breath and respiratory failure). HRCT was considered effective if the patient had received HRCT in the same hospital within 12 months and screening HRCT is not necessary.

  3. Having daily expectoration(with sufficient sputum production at screening, if the subject is unable to produce sputum voluntarily, sample collection can be performed by induced expectoration).

  4. Have at least 2 pulmonary exacerbations in the past 12 months before Screening.

  5. If long-term treatment with bronchodilators (long-acting β-agonists and/or long-acting muscarinic antagonists) is required, the dose and regimen should remain stable for at least 3 months before the screening visit and throughout the study period.

  6. The estimated survival time ≥ 12 months.

  7. Women must be post-menopausal, surgically sterile, or using highly effective contraception methods from Day 1 to at least 30 days after the last dose.

  8. Males with female partners of childbearing potential must be using effective contraception from Day 1 to at least 90 days after the last dose.

  9. Give their signed study informed consent to participate.

Exclusion Criteria:

* 1. Have pulmonary hypertension or have a primary diagnosis of COPD or asthma as judged by the Investigator.

  2. A history of malignancy (excluding cured basal cell carcinoma of the skin, carcinoma in situ, and papillary carcinoma of the thyroid gland. The patients who had survived lung cancer surgery for at least 5 years without antitumor therapy can enroll in the study ) within 5 years prior to screening or a history of antitumor therapy.

  3. Have bronchiectasis due to CF (HRCT showed that the above lung diseases became predominant) as judged by the Investigator.

  4. Currently being treated Non-tuberculous Mycobacterial (NTM) pulmonary infections, allergic bronchopulmonary aspergillosis, or tuberculosis (TB), or active and currently symptomatic infections caused by COVID-19.

  5. Patients who had experienced any degree of acute exacerbation of bronchiectasis or were developing an acute exacerbation of bronchiectasis before 4 weeks of screening.

  6. Patients who had hemoptysis and required medical intervention within 4 weeks prior to screening(except for coughing up minorbloody streaks).

  7. Have an abnormal renal function test result (estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73m^2) at Screening.

  8. Subjects with a history of liver disease or current treatment for liver disease during the screening period, including but not limited to acute or chronic hepatitis, cirrhosis or liver failure, or aspartate aminotransferase (AST) > 2.0×ULN or alanine aminotransferase (ALT) > 2.0×ULN or total bilirubin (TBIL) > 1.5×ULN.

  9. Active hepatitis B virus infection (hepatitis B surface antigen positive with HBV-DNA load above the lower limit of detection), active hepatitis C virus infection (HCV antibody positive with HCV-RNA load above the lower limit of detection), or known HIV infection or syphilis infection.

  10. Any other unstable clinical condition, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematologic, psychiatric, or major physiological dysfunction, that the investigator considers to be (a) likely to affect patient safety throughout the study; (b) Influence the results of the study and its interpretation; (c) impeding the patient's ability to complete the entire study.

  11. Had participated in a clinical trial of any other drug or medical device in the 3 months prior to the screening (a drug or medical device treated with a clinical trial) or the subject had not been more than 5 half-lives from the last clinical trial of the drug at the time of screening.

  12. Medications that may cause hyperkeratosis (e.g., tumor necrosis factor-α antagonists) within 4 weeks prior to screening.

  13. Patients who have used a strong inducer or suppressor of CYP3A within 14 days or 5 half-lives of the first investigational drug (whichever is longer).

  14. Patients who had smoked an average of 10 cigarettes or more per day in the previous 1 year were screened.

  15. Pregnancy and lactation.

  16. The subjects were unable to complete the questionnaires due to their limited educational level, or the subjects and their families failed to fill in the subjects' log cards.

  17. Had received live attenuated vaccine within 30 days before randomization. 18. The investigators judged that there were other conditions that were not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Frequency of pulmonary exacerbations | 24-week treatment period
  Number of events per person-time over 24-weeks

SECONDARY OUTCOMES:
Time to first pulmonary exacerbation | 24-week treatment period
  Exacerbation is defined by signs and symptoms plus intervention with systemic antibiotics
Change from Baseline(Screening) in forced expiratory volume in 1 second (FEV1) | 24-week treatment period
  Change from Baseline(Screening) in FEV1 at 24-weeks
Change from Baseline(Screening) in 24-hour Sputum Weight and Sputum purulence score | 24-week treatment period
  Change from Baseline(Screening) in 24h Sputum Weight and Purulence Score at 24-weeks
Change from Baseline(Screening) in Frequency of Hemoptysis | 24-week treatment period
  Change from Baseline(Screening) in Hemoptysis
Change from Baseline in the Respiratory Symptoms Domain Score of the Quality of Life (QOL) Bronchiectasis questionnaire | 24-week treatment period
  Change from Baseline Quality of Life (QOL) Bronchiectasis questionnairescore at 24-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Weijie Guan, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker AF. Bronchiectasis. N Engl J Med. 2002 May 2;346(18):1383-93. doi: 10.1056/NEJMra012519. No abstract available. PMID 11986413
- [Background] Chalmers JD, Aliberti S, Filonenko A, Shteinberg M, Goeminne PC, Hill AT, Fardon TC, Obradovic D, Gerlinger C, Sotgiu G, Operschall E, Rutherford RM, Dimakou K, Polverino E, De Soyza A, McDonnell MJ. Characterization of the "Frequent Exacerbator Phenotype" in Bronchiectasis. Am J Respir Crit Care Med. 2018 Jun 1;197(11):1410-1420. doi: 10.1164/rccm.201711-2202OC. PMID 29357265
- [Derived] Zhong NS, Qiu R, Cao J, Huang YM, Zhou H, Xu XX, Xu JF, Ye H, Yang ZR, Gao LY, Shen Y, Xiao ZK, Xie SG, Lin DJ, Zhao L, Xiong H, Zhang XM, Li FQ, Guan WJ, Chalmers JD; SAVE-BE trial investigators. Effects of the DPP-1 inhibitor HSK31858 in adults with bronchiectasis in China (SAVE-BE): a phase 2, multicentre, double-blind, randomised, placebo-controlled trial. Lancet Respir Med. 2025 May;13(5):414-424. doi: 10.1016/S2213-2600(25)00019-0. Epub 2025 Mar 25. PMID 40154523
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11986413/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29357265/